CLINICAL TRIAL: NCT00104312
Title: Weakness From Inflammation: A Basis of Disability From Knee Osteoarthritis
Brief Title: Osteoarthritis: Weakness From Inflammation
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Shari Ling, MD, Principal Investigator, National Institute on Aging
Other Study IDs: AG0016
Record Dates: First submitted 2005-02-24; First posted 2005-02-25 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Osteoarthritis
Keywords: Knee Osteoarthritis; Muscle; Cytokine; Mobility; Function
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Synovial fluid and tissue blood serum muscle biopsy

GROUPS / COHORTS (2):
- 1: Participants with symptomatic knee osteoarthritis
- 2: Participants without symptomatic knee osteoarthritis, age-matched as controls

SUMMARY:
The purpose of this study is to understand the factors that lead to muscle weakness with arthritis and aging.

DETAILED DESCRIPTION:
Through this study, we hope to learn about the natural history of knee osteoarthritis and the disability that arises from it. We hope to better understand why people with knee osteoarthritis develop difficulty with mobility (e.g. walking, standing) in hopes of finding a cure.

This study requires 1 four-hour visit to Harbor Hospital. The visit involves a physical exam, a DEXA bone density scan, blood and urine testing, knee x-rays, strength testing and a surface electromyography (EMG). Samples of muscle, joint fluid and joint tissue will be collected during your planned surgery.

Participation in this study is entirely voluntary.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* Normal body weight (a Body Mass Index (BMI) of 30 or less)
* Osteoarthritis of the knee (prior to knee surgery)
* Planning to have knee surgery at a MedStar Hospital

Exclusion Criteria:

* History of a stroke
* History of muscle weakness or paralysis
* History of Rheumatoid Arthritis or
* Inflammatory Joint Disease
* History of a Bleeding Disorder
* History of Gout
* Diabetes for which you take insulin
* Polymyalgia rheumatica (total body muscle aching/stiffness)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community - Men and women
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2001-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shari Ling, MD, Principal Investigator — NIA, Johns Hopkins Medical Institution Divisions of Rheumatology, Gerontology, and Geriatrics
Locations (1):
- Harbor Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Cooper C, Snow S, McAlindon TE, Kellingray S, Stuart B, Coggon D, Dieppe PA. Risk factors for the incidence and progression of radiographic knee osteoarthritis. Arthritis Rheum. 2000 May;43(5):995-1000. doi: 10.1002/1529-0131(200005)43:53.0.CO;2-1. PMID 10817551
- [Background] Slemenda C, Heilman DK, Brandt KD, Katz BP, Mazzuca SA, Braunstein EM, Byrd D. Reduced quadriceps strength relative to body weight: a risk factor for knee osteoarthritis in women? Arthritis Rheum. 1998 Nov;41(11):1951-9. doi: 10.1002/1529-0131(199811)41:113.0.CO;2-9. PMID 9811049
- [Background] Conwit RA, Stashuk D, Tracy B, McHugh M, Brown WF, Metter EJ. The relationship of motor unit size, firing rate and force. Clin Neurophysiol. 1999 Jul;110(7):1270-5. doi: 10.1016/s1388-2457(99)00054-1. PMID 10423192